CLINICAL TRIAL: NCT01933971
Title: Evaluation of Dose-response, Pharmacodynamic and Pharmacokinetic Bioequivalence of Filgrastim in Healthy Male Volunteers After Single and Multiple-dose Subcutaneous Administration of the BK0023 Injectable Formulation vs. Neupogen®
Brief Title: Evaluation of Dose-response, Pharmacodynamic and Pharmacokinetic Bioequivalence of Filgrastim in Healthy Male Volunteers After Single and Multiple-dose Subcutaneous Administration of the Test Injectable Formulation BK0023 vs. Neupogen®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-ker S.r.l. (Industry)
Collaborators: Cross Research S.A. (Industry); Nerviano Medical Sciences (Industry); AAI Deutschland GmbH & Co. KG (Other); Gife S.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-PK-06-175; 2007DR1116 (Other: Swissmedic)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: filgrastim 2.5 µg/kg/day for 7 consecutive days (Other): The test investigational product is BK0023. The reference product is Neupogen® 30, by Dompé Biotec S.p.A., Italy.
  Both study treatments were administered according to a cross-over design in 2 subsequent periods separated by wash-out periods of at least 28 days.
  The sites, where the injections are to be performed, are planned as follows:
  1. st injection: upper part of the upper arm, posterior surface
  2. nd injection: upper part of the thigh
  3. rd injection: abdomen with the exception of the umbilical area
  4. th injection: upper part of the contra-lateral upper arm, posterior surface
  5. th injection: upper part of the contra-lateral thigh
  6. th injection: abdomen with the exception of the umbilical area
  7. th injection: upper part of the same upper arm, posterior surface as for the 1st injection.
  Interventions: Drug: Filgrastim test; Drug: Filgrastim reference
- Group 2: filgrastim 5 µg/kg/day for 7 consecutive days (Other): The test investigational product is BK0023. The reference product is Neupogen® 30, by Dompé Biotec S.p.A., Italy.
  Both study treatments were administered according to a cross-over design in 2 subsequent periods separated by wash-out periods of at least 28 days.
  The sites, where the injections are to be performed, are planned as follows:
  1. st injection: upper part of the upper arm, posterior surface
  2. nd injection: upper part of the thigh
  3. rd injection: abdomen with the exception of the umbilical area
  4. th injection: upper part of the contra-lateral upper arm, posterior surface
  5. th injection: upper part of the contra-lateral thigh
  6. th injection: abdomen with the exception of the umbilical area
  7. th injection: upper part of the same upper arm, posterior surface as for the 1st injection.
  Interventions: Drug: Filgrastim test; Drug: Filgrastim reference
- Group 3: filgrastim 10 µg/kg/day for 5 consecutive days (Other): The test investigational product is BK0023. The reference product is Neupogen® 30, by Dompé Biotec S.p.A., Italy.
  Both study treatments were administered according to a cross-over design in 2 subsequent periods separated by wash-out periods of at least 28 days.
  The sites, where the injections are to be performed, are planned as follows:
  1. st injection: upper part of the upper arm, posterior surface
  2. nd injection: upper part of the thigh
  3. rd injection: abdomen with the exception of the umbilical area
  4. th injection: upper part of the contra-lateral upper arm, posterior surface
  5. th injection: upper part of the contra-lateral thigh.
  Interventions: Drug: Filgrastim test; Drug: Filgrastim reference

INTERVENTIONS:
Drug: Filgrastim test — 0.3 mg/mL injectable solution in 1 mL vials Manufacturer (Drug Substance): Eurogenetec S.A., B-4102 Seraing, Belgium Manufacturer (Drug Product): Areta International S.r.l., I-21040 Gerenzano, Italy Batch release: Areta International S.r.l., I-21040 Gerenzano, Italy Route of administration: subcutaneous
  Other Names: r-metHuG-CSF, BK0023
Drug: Filgrastim reference — 0.3 mg/mL injectable solution in 1 mL vials Licensed owner: Dompé farmaceutici S.p.A., Milan, Italy Manufacturer (Drug Product): Hoffmann - La Roche Ltd., Basel, Switzerland and Amgen Manufacturing Limited, Puertorico.
  Batch release: Amgen Europe B.V., Breda, Netherlands Route of administration: subcutaneous
  Other Names: r-metHuG-CSF, Neupogen®

SUMMARY:
Study rationale: Bio-ker has developed the new formulation of filgrastim BK0023 with the same active content as Neupogen®. BK0023 is expected to have the same tolerability profile and clinical effects as Neupogen® in controlling myelo-toxicity induced by chemotherapy given for the treatment of solid and haematological tumours. It is worth noting that the production and manufacturing procedures allow to have a reduction of drug cost thus it is likely to have pharmacoeconomic advantages.

The study is aimed at investigating the pharmacodynamic equivalence and the pharmacokinetic bioequivalence of the new BK0023 injectable formulation of filgrastim 0.3 mg/mL by Bio-Ker S.r.l. vs. the comparator (Neupogen® 0.3 mg/mL, Dompé Biotec S.p.A., Italy). Healthy male subjects will receive test and reference at the doses of 2.5 and 5 µg/kg/day for 7 consecutive days and at the dose of 10 µg/kg/day for 5 consecutive days according to a randomised cross-over design. Pharmacodynamics, pharmacokinetics and safety of BK0023 injectable formulation 0.3 mg/mL and of Neupogen® 0.3 mg/mL, administered in 2 consecutive periods with a wash-out of at least 28 days elapsing between the last injection of period I and the first of period II, are compared.

Study design: Single and multiple escalating dose, double-blind, randomised, two-way cross-over, pharmacodynamic and pharmacokinetic bioequivalence study.

DETAILED DESCRIPTION:
In a first part of the study, 16 healthy male subjects will be included in each dose group and will receive test and reference product according to the cross-over design. After the end of the second period of each dose group (completion of both cross-over periods for each dose group) the pharmacodynamic and pharmacokinetic primary parameters will be calculated. The blinding will be temporarily broken by one statistician for the ad interim analysis of primary parameters that will be performed after conclusion of the treatment of 16 subjects for each dose group (results are not disclosed) with the aim to re-calculate the sample size and to conclude the study with the necessary and sufficient number of subjects for each dose regimen.

The study design was chosen according to the internationally recognised guideline for pharmacokinetics studies and in accordance with the EMEA guidance on similar medicinal products containing recombinant granulocyte-colony stimulating factor (G-CSF), which is annexed to the guideline on similar biological medicinal products containing biotechnology-derived proteins as active substance: non-clinical and clinical issues. A clinical development plan including the study outline was also submitted to EMEA, which examined the documentation and gave advice about the present study design .

A multiple-dose design was chosen instead of a single-dose design, since G-CSF pharmacokinetics is non linear due to 2 reasons: non-proportional increase with dose and time dependent non-linearity. However, pharmacodynamic equivalence and pharmacokinetic bioequivalence will be both tested after the 1st and the last dose of the multiple dose treatment.

Since the effects of r-h-met-G-CSF can be directly measured as pharmacodynamic responses, i.e. the increase in the absolute neutrophil count (ANC) and the development of peripheral blood cells (CD34+ cells), both parameters will be evaluated for the equivalence testing.

Dose levels of 2.5 and 5 μg/kg/day were chosen for the pharmacodynamic equivalence, since literature data show a clear dose-response relationship in terms of the pharmacodynamic parameters over this range. The 10 μg/kg/day dose was chosen to make the investigated range relevant with respect to the clinical indications and the usual praxis for Neupogen®. Moreover, the subcutaneous administration was chosen, since this administration route is the most commonly used in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* a body mass index (BMI) between 18 and 28 kg/m2,
* a body weight between 60 and 90 kg,
* good health based on medical history, physical examination, a 12-lead electrocardiogram (ECG) and routine haematology and blood chemistry tests,
* willingness to provide written informed consent
* values of leukocytes and thrombocytes had to be inside the normality range at the screening.

Exclusion Criteria:

* intake of any concomitant medication,
* a history of drug, caffeine (>5 cups coffee/tea/day) or tobacco (>/=10 cigarettes/day) abuse, or alcohol consumption in excess of two drinks per day, as defined by the U.S.D.A. dietary guidelines,
* ascertained or presumptive hypersensitivity to the active compound or history of anaphylaxis to drugs.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve of absolute neutrophil count (AUCANCday1) and maximum absolute neutrophil count (ANCday1max); AUCANCday1-10 and AUCANCday1-8; ANCday1-10max and ANCday1-8max; AUCday1 and AUCss of filgrastim in serum. | Day 1 after single dose and from day 1 to 10 (dose groups of 2.5 and 5 µg/kg/day) or from day 1 to 8 (dose group of 10 µg/kg/day)
  Baseline adjusted AUC of ANC on day 1 after single dose (AUCANCday1) and from day 1 to 10 (dose groups of 2.5 and 5 µg/kg/day) or from day 1 to 8 (dose group of 10 µg/kg/day) including the elimination period (AUCANCday1-10 and AUCANCday1-8) and ANCday1max, ANCday1-10max and ANCday1-8max after treatment with filgrastim 0.3 mg/mL by Bio-ker and Neupogen® AUC of serum filgrastim after both single (AUCday1) and multiple dose (AUCss) of filgrastim 0.3 mg/mL by Bio-ker and Neupogen®

SECONDARY OUTCOMES:
Area under the curve of CD34+ cell count (AUCCD34+) and maximum CD34+ cell count (CD34+max); maximum concentrations at steady state (Cssmax), Cmaxday1, time to achieve Cmax (Tmax), t1/2 and clearance of serum filgrastim | On day 1 after single dose and from day 1 to 10 (dose groups of 2.5 and 5 µg/kg/day) or from day 1 to 8 (dose group of 10 µg/kg/day)
  Baseline adjusted AUCCD34+ from day 1 to 10 (dose groups of 2.5 and 5 µg/kg/day) or from day 1 to 8 (dose group of 10 µg/kg/day) including the elimination period and CD34+max after treatment with filgrastim 0.3 mg/mL by Bio-ker and Neupogen® Cmax, Tmax t1/2 and clearance of serum filgrastim after both single (Cmaxday1, Tmaxday1, t1/2day1 and Clday1) and multiple dose (Cssmax, Tssmax, tss1/2, Clss) of filgrastim 0.3 mg/mL by Bio-ker and Neupogen®

OTHER OUTCOMES:
adverse events, blood pressure, heart rate, body temperature, body weight, ECGs, clinical laboratory assays | From day 1 to 10 (dose groups of 2.5 and 5 µg/kg/day) or from day 1 to 8 (dose group of 10 µg/kg/day)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Rusca, MD, Principal Investigator — CROSS Research SA
Locations (1):
- CROSS Research SA, Arzo, Canton Ticino, Switzerland

REFERENCES:
- [Background] Hryniuk W, Bush H. The importance of dose intensity in chemotherapy of metastatic breast cancer. J Clin Oncol. 1984 Nov;2(11):1281-8. doi: 10.1200/JCO.1984.2.11.1281. No abstract available. PMID 6387060
- [Background] Gardner SN. A mechanistic, predictive model of dose-response curves for cell cycle phase-specific and -nonspecific drugs. Cancer Res. 2000 Mar 1;60(5):1417-25. PMID 10728708
- [Background] Skipper HE. Kinetics of mammary tumor cell growth and implications for therapy. Cancer. 1971 Dec;28(6):1479-99. doi: 10.1002/1097-0142(197112)28:63.0.co;2-m. No abstract available. PMID 5127796
- [Background] Skipper HE, Schabel FM, Lloyd HH. Dose-response and tumour cell repopulation rate in chemotherapeutic trials. Adv Cancer Chemother 1: 205-253, 1979
- [Background] Welte K, Platzer E, Lu L, Gabrilove JL, Levi E, Mertelsmann R, Moore MA. Purification and biochemical characterization of human pluripotent hematopoietic colony-stimulating factor. Proc Natl Acad Sci U S A. 1985 Mar;82(5):1526-30. doi: 10.1073/pnas.82.5.1526. PMID 3871951
- [Background] Nomura H, Imazeki I, Oheda M, Kubota N, Tamura M, Ono M, Ueyama Y, Asano S. Purification and characterization of human granulocyte colony-stimulating factor (G-CSF). EMBO J. 1986 May;5(5):871-6. doi: 10.1002/j.1460-2075.1986.tb04297.x. PMID 3487449
- [Background] Simmers RN, Webber LM, Shannon MF, Garson OM, Wong G, Vadas MA, Sutherland GR. Localization of the G-CSF gene on chromosome 17 proximal to the breakpoint in the t(15;17) in acute promyelocytic leukemia. Blood. 1987 Jul;70(1):330-2. PMID 2439153
- [Background] Nicola NA. Hemopoietic cell growth factors and their receptors. Annu Rev Biochem. 1989;58:45-77. doi: 10.1146/annurev.bi.58.070189.000401. No abstract available. PMID 2549855
- [Background] Nicola NA, Metcalf D, Matsumoto M, Johnson GR. Purification of a factor inducing differentiation in murine myelomonocytic leukemia cells. Identification as granulocyte colony-stimulating factor. J Biol Chem. 1983 Jul 25;258(14):9017-23. PMID 6190815
- [Background] Nicola NA, Begley CG, Metcalf D. Identification of the human analogue of a regulator that induces differentiation in murine leukaemic cells. Nature. 1985 Apr 18-24;314(6012):625-8. doi: 10.1038/314625a0. PMID 2986009
- [Background] Fukunaga R, Ishizaka-Ikeda E, Nagata S. Purification and characterization of the receptor for murine granulocyte colony-stimulating factor. J Biol Chem. 1990 Aug 15;265(23):14008-15. PMID 1696260
- [Background] Layton JE, Hall NE, Connell F, Venhorst J, Treutlein HR. Identification of ligand-binding site III on the immunoglobulin-like domain of the granulocyte colony-stimulating factor receptor. J Biol Chem. 2001 Sep 28;276(39):36779-87. doi: 10.1074/jbc.M104787200. Epub 2001 Jul 23. PMID 11468284
- [Background] Shimoda K, Okamura S, Harada N, Kondo S, Okamura T, Niho Y. Identification of a functional receptor for granulocyte colony-stimulating factor on platelets. J Clin Invest. 1993 Apr;91(4):1310-3. doi: 10.1172/JCI116330. PMID 7682568
- [Background] Boneberg EM, Hareng L, Gantner F, Wendel A, Hartung T. Human monocytes express functional receptors for granulocyte colony-stimulating factor that mediate suppression of monokines and interferon-gamma. Blood. 2000 Jan 1;95(1):270-6. PMID 10607712
- [Background] Bussolino F, Wang JM, Defilippi P, Turrini F, Sanavio F, Edgell CJ, Aglietta M, Arese P, Mantovani A. Granulocyte- and granulocyte-macrophage-colony stimulating factors induce human endothelial cells to migrate and proliferate. Nature. 1989 Feb 2;337(6206):471-3. doi: 10.1038/337471a0. PMID 2464767
- [Background] Souza LM, Boone TC, Gabrilove J, Lai PH, Zsebo KM, Murdock DC, Chazin VR, Bruszewski J, Lu H, Chen KK, Barendt J, Platzer E, Moore MAS, Mertelsmann R, Welte K. Recombinant human granulocyte colony-stimulating factor: effects on normal and leukemic myeloid cells. Science. 1986 Apr 4;232(4746):61-5. doi: 10.1126/science.2420009.
- [Background] Zsebo KM, Cohen AM, Murdock DC, Boone TC, Inoue H, Chazin VR, Hines D, Souza LM. Recombinant human granulocyte colony stimulating factor: molecular and biological characterization. Immunobiology. 1986 Sep;172(3-5):175-84. doi: 10.1016/S0171-2985(86)80097-3. PMID 3492428
- [Background] Bonig H, Silbermann S, Weller S, Kirschke R, Korholz D, Janssen G, Gobel U, Nurnberger W. Glycosylated vs non-glycosylated granulocyte colony-stimulating factor (G-CSF)--results of a prospective randomised monocentre study. Bone Marrow Transplant. 2001 Aug;28(3):259-64. doi: 10.1038/sj.bmt.1703136. PMID 11535993
- [Background] Gabrilove JL, Jakubowski A, Scher H, Sternberg C, Wong G, Grous J, Yagoda A, Fain K, Moore MA, Clarkson B, Oettgen HF, Alton K, Welte K, Souza L. Effect of granulocyte colony-stimulating factor on neutropenia and associated morbidity due to chemotherapy for transitional-cell carcinoma of the urothelium. N Engl J Med. 1988 Jun 2;318(22):1414-22. doi: 10.1056/NEJM198806023182202. PMID 2452983
- [Background] Glaspy JA, Baldwin GC, Robertson PA, Souza L, Vincent M, Ambersley J, Golde DW. Therapy for neutropenia in hairy cell leukemia with recombinant human granulocyte colony-stimulating factor. Ann Intern Med. 1988 Nov 15;109(10):789-95. doi: 10.7326/0003-4819-109-10-789. PMID 2461131
- [Background] Fabian I, Kletter Y, Bleiberg I, Gadish M, Naparsteck E, Slavin S. Effect of exogenous recombinant human granulocyte and granulocyte-macrophage colony-stimulating factor on neutrophil function following allogeneic bone marrow transplantation. Exp Hematol. 1991 Oct;19(9):868-73. PMID 1716591
- [Background] Welte K, Gabrilove J, Bronchud MH, Platzer E, Morstyn G. Filgrastim (r-metHuG-CSF): the first 10 years. Blood. 1996 Sep 15;88(6):1907-29. No abstract available. PMID 8822908
- [Background] Morstyn G, Campbell L, Souza LM, Alton NK, Keech J, Green M, Sheridan W, Metcalf D, Fox R. Effect of granulocyte colony stimulating factor on neutropenia induced by cytotoxic chemotherapy. Lancet. 1988 Mar 26;1(8587):667-72. doi: 10.1016/s0140-6736(88)91475-4. PMID 2895212
- [Background] Crawford J, Ozer H, Stoller R, Johnson D, Lyman G, Tabbara I, Kris M, Grous J, Picozzi V, Rausch G, et al. Reduction by granulocyte colony-stimulating factor of fever and neutropenia induced by chemotherapy in patients with small-cell lung cancer. N Engl J Med. 1991 Jul 18;325(3):164-70. doi: 10.1056/NEJM199107183250305. PMID 1711156
- [Background] Pettengell R, Gurney H, Radford JA, Deakin DP, James R, Wilkinson PM, Kane K, Bentley J, Crowther D. Granulocyte colony-stimulating factor to prevent dose-limiting neutropenia in non-Hodgkin's lymphoma: a randomized controlled trial. Blood. 1992 Sep 15;80(6):1430-6. PMID 1381626
- [Background] Trillet-Lenoir V, Green J, Manegold C, Von Pawel J, Gatzemeier U, Lebeau B, Depierre A, Johnson P, Decoster G, Tomita D, et al. Recombinant granulocyte colony stimulating factor reduces the infectious complications of cytotoxic chemotherapy. Eur J Cancer. 1993;29A(3):319-24. doi: 10.1016/0959-8049(93)90376-q. PMID 7691119
- [Background] Maher DW, Lieschke GJ, Green M, Bishop J, Stuart-Harris R, Wolf M, Sheridan WP, Kefford RF, Cebon J, Olver I, McKendrick J, Toner G, Bradstock K, Lieschke M, Cruickshank S, Tomita DK, Hoffman EW, Fox RM, Morstyn G. Filgrastim in patients with chemotherapy-induced febrile neutropenia. A double-blind, placebo-controlled trial. Ann Intern Med. 1994 Oct 1;121(7):492-501. doi: 10.7326/0003-4819-121-7-199410010-00004. PMID 7520676
- [Background] Vial T, Descotes J. Clinical toxicity of cytokines used as haemopoietic growth factors. Drug Saf. 1995 Dec;13(6):371-406. doi: 10.2165/00002018-199513060-00006. PMID 8652081
- [Background] Lindemann A, Herrmann F, Oster W, Haffner G, Meyenburg W, Souza LM, Mertelsmann R. Hematologic effects of recombinant human granulocyte colony-stimulating factor in patients with malignancy. Blood. 1989 Dec;74(8):2644-51. PMID 2479425
- [Background] Sakamaki S, Matsunaga T, Hirayama Y, Kuga T, Niitsu Y. Haematological study of healthy volunteers 5 years after G-CSF. Lancet. 1995 Nov 25;346(8987):1432-3. doi: 10.1016/s0140-6736(95)92450-7. No abstract available. PMID 7475852
- [Background] Borleffs JC, Bosschaert M, Vrehen HM, Schneider MM, van Strijp J, Small MK, Borkett KM. Effect of escalating doses of recombinant human granulocyte colony-stimulating factor (filgrastim) on circulating neutrophils in healthy subjects. Clin Ther. 1998 Jul-Aug;20(4):722-36. doi: 10.1016/s0149-2918(98)80135-5. PMID 9737832
- [Background] Note for Guidance on the Investigation of Bioavailability and Bioequivalence, The European Agency for the Evaluation of Medicinal Products (EMEA), guideline CPMP/EWP/QWP/1401/98, London, 26 July 2001
- [Background] Annex guideline on similar biological medicinal products containing biotechnology-derived proteins as active substance: non-clinical and clinical issues,
- [Background] Tanaka R, Matsudaira T, Aizawa J, Ebihara Y, Muraoka K, Tsuji K, Ikebuchi K, Kodama K, Takaku F, Nakahata T. Characterization of peripheral blood progenitor cells (PBPC) mobilized by filgrastim (rHuG-CSF) in normal volunteers: dose-effect relationship for filgrastim with the character of mobilized PBPC. Br J Haematol. 1996 Mar;92(4):795-803. doi: 10.1046/j.1365-2141.1996.412949.x. PMID 8616069
- [Background] Chow S and J Liu (2000), Design and analysis of bioavailability and bioequivalence studies, 2nd Edition, Revised and expanded, Marcel Dekker Inc., New York - Basel.
- [Background] van Der Auwera P, Platzer E, Xu ZX, Schulz R, Feugeas O, Capdeville R, Edwards DJ. Pharmacodynamics and pharmacokinetics of single doses of subcutaneous pegylated human G-CSF mutant (Ro 25-8315) in healthy volunteers: comparison with single and multiple daily doses of filgrastim. Am J Hematol. 2001 Apr;66(4):245-51. doi: 10.1002/ajh.1052. PMID 11279634
- [Background] Houston AC, Stevens LA, Cour V. Pharmacokinetics of glycosylated recombinant human granulocyte colony-stimulating factor (lenograstim) in healthy male volunteers. Br J Clin Pharmacol. 1999 Mar;47(3):279-84. doi: 10.1046/j.1365-2125.1999.00888.x. PMID 10215752
- [Background] Hoglund M, Smedmyr B, Bengtsson M, Totterman TH, Cour-Chabernaud V, Yver A, Simonsson B. Mobilization of CD34+ cells by glycosylated and nonglycosylated G-CSF in healthy volunteers--a comparative study. Eur J Haematol. 1997 Sep;59(3):177-83. doi: 10.1111/j.1600-0609.1997.tb00972.x. PMID 9310126
- [Background] U.S. Department of Health and Human Services and U.S. Department of Agriculture, Nutrition and your health: Dietary Guidelines for Americans, 2005
- [Derived] Crobu D, Spinetti G, Schrepfer R, Tonon G, Jotti GS, Onali P, Dedoni S, Orsini G, Di Stefano A. Preclinical and clinical phase I studies of a new recombinant Filgrastim (BK0023) in comparison with Neupogen(R). BMC Pharmacol Toxicol. 2014 Feb 21;15:7. doi: 10.1186/2050-6511-15-7. PMID 24555723